CLINICAL TRIAL: NCT04107610
Title: Development of a Pediatric Oculomotor and Vestibular Normative Database as an Essential Tool for Objective Evaluation of Concussion and Return-to-school/Play
Brief Title: Normative Oculomotor and Vestibular Data in Pediatric Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neurolign (Industry)
Collaborators: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pediatric SBIR
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: oculomotor,; vestibular,; concussion,; mild traumatic brain injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: I-PAS — I-PAS is a portable, head-mounted display goggle system with integrated eye tracking technology. I-PAS records eye movements in response to visual and auditory stimuli.

SUMMARY:
The purpose of this study is to use a device called I-Portal® Portable Assessment System (I-PAS) to record eye movements in response to a number of visual and auditory stimuli designed to evaluate neural brain pathways related to oculomotor, vestibular, reaction time and cognitive (OVRT-C) development. The goal of this research is to collect normative data for the OVRT-C tests from a healthy pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 6 to 18 years of all races.
* Parental/guardian permission (informed consent) and child assent

Exclusion Criteria:

* History of head injury characterized by any of the following:

  1. Resulting from penetrating trauma
  2. Resulting from an automobile accident with significant associated injuries
  3. Associated with a Glasgow Comma Scale Score of less than 13 at the time of injury
  4. Associated with a loss of consciousness period greater than 30 minutes
  5. Judged to be more than mild by medical staff
  6. Requiring admission to the hospital for any reason
  7. Associated with subdural or epidural hemorrhage
  8. Persons with a previous history of mTBI in the past and who were symptomatic prior to current injury
* Pregnancy, as documented by last menstrual period at study visits
* Implants: Persons implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant, metal cervical spine hardware
* Diagnosed with attention deficit hyperactivity disorder (ADHD), autism spectrum disorder, major depression, hypochondriasis, bipolar disorders, or schizophrenia.
* Presence of severe aphasia or inability to follow commands and give independent responses
* Documented neurodegenerative disorders (Multiple sclerosis, Parkinson's, Alzheimer's, Huntington)
* Past history of seizures or convulsions
* Prior disorders of hearing and balance including:

  1. Meniere's disease
  2. Multiple sclerosis
  3. Vestibular neuritis
  4. Vestibular schwannoma
  5. Sudden sensorineural hearing loss
  6. History of ear operation other than myringotomy and tube placement in the past
  7. Acute or chronic disease of middle ear (infections, otitis)
* History of cerebrovascular disorders including stroke, brainstem or cerebellar dysfunction within the last 3 months
* Systemic disorders that include chronic renal failure, cirrhosis of the liver, autoimmune disease, heart disease, lung disease, severe arthritis, diabetes, hypertension
* Repeated history of syncope
* Past or concomitant treatment with ototoxic chemotherapy
* Previous contraindicating surgeries at the discretion of the study physician
* Aminoglycosides in the past 6 months given via systemic or transtympanic administration
* Concomitant treatment with any of the followings within the last 24 hours prior to testing if more than 2 doses have been taken:

  1. Antihistamines: e.g. diphenhydramine, cyclizine, dimenhydrinate, meclizine, hydroxyzine, promethazine,
  2. For ADHD and narcolepsy: e.g. Concerta, Daytrana, Methylin, Ritalin, Ritalin LA, Metadate ER, Aptensio XR, Cotempla XR-ODT, QuilliChew ER, and Quillivant XR
  3. For schizophrenia and other mental diseases: e.g. Phenothiazines
  4. Specific antibiotics: e.g. ethambutol, gentamycin
  5. Anticonvulsant medications: e.g. topiramate
* Currently suffering from dehydration
* History or suspicion of substance abuse or addiction
* Acute alcohol intoxication
* Playing professional sports at the Olympic/league level

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Normative data for I-PAS tests | 3 years
  Accuracy and gain across age: measurements of eye displacement versus stimulus displacement in saccadic and smooth pursuit tasks

SECONDARY OUTCOMES:
Goggle evaluation | 3 years
  Short questionnaire consisting of 6 questions to assess the look, feel and weight of the goggles. 5 questions are Yes/No (0/1) and one question is on a rating from 0 to 3. The total score from these questions represents an evaluation of goggle comfort. The score can be between 0-8, where a score of 0 is indicative of a very good comfort level and a score of 8 of a low comfort level.

CONTACTS AND LOCATIONS:
Overall Officials: Aura Kullmann, PhD, Principal Investigator — Neuro Kinetics/Neurolign; ALEXANDER D KIDERMAN, PhD, Principal Investigator — Neuro Kinetics/Neurolign
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Allegheny Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No